CLINICAL TRIAL: NCT05333432
Title: Evaluation of a Multimodal Strategy for Early Diagnosis of Men at High Genetic Risk of Prostate Cancer
Acronym: HRPCa-II
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: difficulties in setting up the study within the investigation centers in connection with complex organization
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP210359
Record Dates: First submitted 2022-04-11; First posted 2022-04-19 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Prostate Cancer
Keywords: Urology; Oncogenetics; Radiology
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Injections

STUDY DESIGN:
Intervention Model Description: The study is a non-comparative multicenter prospective cohort. It follows annually two population groups according to their initial panel of PC predisposing genes. Therefore, it is not randomised.The follow-up is the same for all the participants: it is non-comparative.
  Participant is benefiting of a substantial and close medical surveillance during 3 years: each participant undergoes 4 annual mpRMI of which 2 are added by the research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Men at high genetic risk of prostate cancer (Other): Cohort of unaffected men from 40 to 70 years olds with high risk of prostate cancer (PC) defined as being a member from a family that meets hereditary PC criteria or by carrying a mutation of a DNA repair gene or a gene specific to PC.
  Interventions: Procedure: Multiparameric MRI with injection

INTERVENTIONS:
Procedure: Multiparameric MRI with injection — Participants have a prostate multiparametric MRI with gadolinium injection (T2, diffusion and perfusion sequences) every year.
  PIRADS-V2 is used as decisional endpoint, and subjective score LIKERT as secondary analysis.
  To compute sensivity and specificity, we consider LIKERT as suspicious and/or malignant (PIRADS-V2 = 3, 4 or 5) as positive.

SUMMARY:
Inherited predisposition to prostate cancer (PC) has been defined by strict clinical criteria or by genetic profile determined by the presence of a deleterious mutation of deoxyribonucleic acid (DNA) repair genes related to breast/ovarian cancers (such as BRCA2, BRCA1) or by PC specific variants (HOXB13 and 8q24CASC19). But currently, recommendations for management and mitigation of PC risk with early screening just emerge for BRCA2 mutation carriers. Our study compares a PC screening strategy based on an annual prostate specific antigen (PSA) test and a clinical examination to a strategy that also includes an annual multiparametric magnetic resonance imaging (mpMRI). It focus not only on 440 unaffected men carrying the BRCA2 mutation, but also on 440 unaffected men member of hereditary PC families with an unidentified mutation or carriers of a mutation of another gene that predisposes to PC, for a total number of participants included of 880. This project estimates the benefits and inconveniences to extend the proposed early diagnosis procedure from unaffected men with BRCA2 mutation to all unaffected men meeting criteria of an inherited predisposition. It should allow to diagnose PC at a more curable stage, and to establish national recommendations for the management of men with high genetic risk of PC useful in clinical routine, depending on typology of the genetic risk. This project aims to efficiently diagnose them, without performing unnecessary biopsies, at curable stage of the disease. It should reduce their risk of death from this cancer known to be of bad prognosis at an advanced stage.

DETAILED DESCRIPTION:
Hereditary prostate cancer (HPC) has been defined by strict clinical criteria and represents 5% of all newly diagnosed prostate cancers (PC). Inherited predisposition to PC is also genetically determined by the presence of a deleterious mutation of DNA repair genes related to breast/ovarian cancers (BRCA2, BRCA1, ATM,...) or of PC specific variants (HOXB13 and 8q24-CASC19).

According typology of genetic risk, predisposition exposes to an earlier age of onset or a more aggressive form of the disease, increasing the risk of death from this cancer.

Currently, abnormal digital rectal examination (DRE) and PSA level above 4ng/mL are validated as an indication for performing a MRI and prostate biopsies to establish PC diagnosis in its frequent sporadic form. Recommendations for the management and the mitigation of PC risk with early screening just emerge for BRCA2 mutation carriers.

The unaffected relatives from these HPC families and the carriers of these mutations are potentially at higher risk of PC and need a dedicated screening procedure.

This project is based on our experience and the results from the international IMPACT study.

Our study will compare this PC screening strategy based on an annual PSA test and a clinical examination to a strategy that also includes an annual multiparametric MRI (mpMRI). Indeed, the PROMIS study has shown that mpMRI is very efficient to detect aggressive PC (sensitivity: 93%), and can identify PC in men with low PSA value. This project will estimate the benefits and inconveniences to extend mpMRI at unaffected men with BRCA2 mutation and potentially to all unaffected men meeting criteria of an inherited predisposition. It should allow to diagnose PC at a more curable stage, and to establish national recommendations for the management of men with high genetic risk of PC useful in clinical routine, depending on typology of the genetic risk.

Indeed, the last French national recommendations (HAS "Haute Autorité de Santé" 2012) in terms of systematic screening for prostate cancer do not include men at high genetic risk. Regarding populations of men at high risk, the HAS indicates that in the current state of knowledge, firstly, identifying the groups of men at higher risk of developing prostate cancer is not in itself sufficient to justify screening; and secondly, that no scientific evidence has been found to justify screening for prostate cancer by assaying PSA in male populations considered to be at higher risk of prostate cancer. But these recommendations were published before the results obtained by the IMPACT study.

The study focuses on 880 unaffected men at high genetic risk of PC: 440 unaffected men carrying the BRCA2 mutation, and also 440 unaffected men member of hereditary PC families with an unidentified mutation or carriers of a mutation of another gene that predisposes to PC.

Participants are pre-screened by the investigators among the files of participants already followed by the urology and/or oncogenetic department. Potential participants of the study have been already identified because they are carrying the BRCA2 mutation or are a member of hereditary PC families with an unidentified mutation or carriers of a mutation of another gene that predisposes to PC. Screened participants are offered to participate to the study by the urologist or the oncogenetic, during a consultation visit which constitutes the inclusion visit.

After the inclusion visit, participants undergo annual follow-up consultation visits, as in standard care, during 3 years.

Each follow-up visit consists of :

* an urologic consultation (clinical examination (DRE) and PSA test)
* a MRI examination The urologic consultation and the MRI examination are scheduled from one year to the next by the urologist.

Radiologists perform MRI, interpret MRI according to the PIRADS-V2 classification and organize the anonymous export of the MRI for centralized review within 15 days of the MRI examination. One of the three referent expert radiologists perform the review of the MRI images, within a week. In case of disagreement between the local and expert interpretations, a third review is performed by one of the two other referent expert radiologists to conclude. In case of disagreement between the 2 expert radiologists, the highest PIRADS-V2 is considered.

In case of abnormal DRE or PSA > 3ng/mL or PIRADS-V2 > 2 on mpMRI, a prostatic biopsy has to be performed as in routine care. The participant continues to be followed by the investigator until the results of biopsy are obtained:

* If PC is diagnosed from biopsies, the referent pathologist of the clinical center makes a standardized report of the pathological analysis of the diagnostic biopsies and organizes anonymous export of scanned slides for centralized review. Two expert pathologists, while blinded to clinical, biological and radiological datas perform the centralized review of positive biopsies at the end of the study. Prostate biopsy pathological analysis are assessed according national referential using International Society of Urological Pathology (ISUP) scoring. The participant then leaves the study prematurely and the date of premature discontinuation is the biopsy date.
* If biopsy is negative, the participant remains enrolled in the study and pursue his annual follow-up.

The result of the study is to be compared to the interim results of the IMPACT study obtained after 3 years of screening (DRE & PSA test) on non affected men carrying or not BRCA2 mutation.

ELIGIBILITY:
Inclusion Criteria:

* Unaffected men at high genetic risk of prostate cancer (PC) defined as being a member from a family that meets hereditary PC criteria or by carrying a mutation of a DNA repair gene (BRCA1 / BRCA2 / CDH1 / MLH1 / MSH2 / MSH6 / PALB2 / PTEN / RAD51C / RAD51D / TP53 / ATM / BARD1 / BLM / BRIP1 / CHEK2 / MRE11A / MLH3 / NBN / RAD50 / STK11) or a gene specific to PC (HOXB13 / 8q24-CASC19)
* Aged between 40 and 70 years old
* Written informed consent signed by the participant
* Affiliated to the social security system

Exclusion Criteria:

* Contraindication for MRI (any foreign metallic bodies: cardiac implantable electronic device (CIED) such as pacemakers, implantable cardioverter defibrillators (ICDs) etc., metallic intraocular foreign bodies, implantable neurostimulation systems, cochlear implants/ear implant, drug infusion pumps (insulin delivery, analgesic drugs, or chemotherapy pumps): If possible, the participant has to remove the device. catheters with metallic components (Swan-Ganz catheter), metallic fragments such as bullets, shotgun pellets, and metal shrapnel , cerebral artery aneurysm clips, magnetic dental implants, tissue expander, artificial limb, hearing aid , piercing, clostrophobia, contrast agents allergy or any other contraindication to contrast agents and to their excipients)
* Treatment with a drug that changes PSA level such as 5 alpha reductase inhibitors (dutastéride, finasteride),
* Prostatic biopsy during the last 2 years, or other progressive cancer or co-morbidities threatening survival at 10 years
* Participant under tutorship or / guardianship, and incapable to give informed consent
* Participation to another interventional clinical trial

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Rate of men diagnosed with PC and aggressive PC (ISUP>3 or T2c-T3) | Through study completion, up to 5 years
  ISUP grade group 2 or higher PC are detected by prostate biopsies which are performed in case of abnormal DRE, PSA > 3ng/mL or PIRADS-V2 > 2 on mpMRI. DRE examination, PSA test and mpMRI examination are annual. Timepoint is at the end of the study.

SECONDARY OUTCOMES:
Rate of men diagnosed with PC according aggressiveness classification (ISUP and TNM) in each genetic group | Through study completion, up to 5 years
  ISUP grade and TNM classification of PC are obtained from prostate biopsies which are performed in case of abnormal DRE, PSA > 3ng/mL or PIRADS-V2 > 2 on mpMRI. DRE examination, PSA test and mpMRI examination are annual. Timepoint is at the end of the study.
Rate of performed prostatic biopsies | Through study completion, up to 5 years
  Prostatic biopsies are performed after each abnormal DRE, PSA > 3ng/ml or PIRADS-V2 > 2 on mpMRI.Timepoint is at the end of the study.
Rate of men diagnosed with PC using mpMRI with or without perfusion sequence | Through study completion, up to 5 years
  Dynamic Contrast Enhanced (DCE) score is obtained with perfusion sequence. mpMRI with PIRADS-V2 = 3 with a positive DCE score is reclassified PIRADS-V2 = 4. Rate of men diagnosed with PC is compared using this reclassification or not.
Rate of men diagnosed with PC according to the type of deleterious mutations, and genetic background/environment modulators of risk | Through study completion, up to 5 years
  Participants are classified according to the type of deleterious mutations and genetic background/environment modulators of risk at the inclusion visit (with the demographics and clinical questionnaires). Rate of men diagnosed with PC is compared in each group.
Rate of adverse events related to the diagnostic procedures | Through study completion, up to 5 years
  Adverse events related to every diagnostic procedures (DRE, PSA, mpMRI and prostate biopsy) are collected during the study

CONTACTS AND LOCATIONS:
Overall Officials: Pierre MONGIAT-ARTUS, PUPH, Study Director — Department of Urology - Hôpital Saint Louis - APHP Sorbonne Université

REFERENCES:
- [Background] Ahmed HU, El-Shater Bosaily A, Brown LC, Gabe R, Kaplan R, Parmar MK, Collaco-Moraes Y, Ward K, Hindley RG, Freeman A, Kirkham AP, Oldroyd R, Parker C, Emberton M; PROMIS study group. Diagnostic accuracy of multi-parametric MRI and TRUS biopsy in prostate cancer (PROMIS): a paired validating confirmatory study. Lancet. 2017 Feb 25;389(10071):815-822. doi: 10.1016/S0140-6736(16)32401-1. Epub 2017 Jan 20. PMID 28110982
- [Background] Page EC, Bancroft EK, Brook MN, Assel M, Hassan Al Battat M, Thomas S, Taylor N, Chamberlain A, Pope J, Raghallaigh HN, Evans DG, Rothwell J, Maehle L, Grindedal EM, James P, Mascarenhas L, McKinley J, Side L, Thomas T, van Asperen C, Vasen H, Kiemeney LA, Ringelberg J, Jensen TD, Osther PJS, Helfand BT, Genova E, Oldenburg RA, Cybulski C, Wokolorczyk D, Ong KR, Huber C, Lam J, Taylor L, Salinas M, Feliubadalo L, Oosterwijk JC, van Zelst-Stams W, Cook J, Rosario DJ, Domchek S, Powers J, Buys S, O'Toole K, Ausems MGEM, Schmutzler RK, Rhiem K, Izatt L, Tripathi V, Teixeira MR, Cardoso M, Foulkes WD, Aprikian A, van Randeraad H, Davidson R, Longmuir M, Ruijs MWG, Helderman van den Enden ATJM, Adank M, Williams R, Andrews L, Murphy DG, Halliday D, Walker L, Liljegren A, Carlsson S, Azzabi A, Jobson I, Morton C, Shackleton K, Snape K, Hanson H, Harris M, Tischkowitz M, Taylor A, Kirk J, Susman R, Chen-Shtoyerman R, Spigelman A, Pachter N, Ahmed M, Ramon Y Cajal T, Zgajnar J, Brewer C, Gadea N, Brady AF, van Os T, Gallagher D, Johannsson O, Donaldson A, Barwell J, Nicolai N, Friedman E, Obeid E, Greenhalgh L, Murthy V, Copakova L, Saya S, McGrath J, Cooke P, Ronlund K, Richardson K, Henderson A, Teo SH, Arun B, Kast K, Dias A, Aaronson NK, Ardern-Jones A, Bangma CH, Castro E, Dearnaley D, Eccles DM, Tricker K, Eyfjord J, Falconer A, Foster C, Gronberg H, Hamdy FC, Stefansdottir V, Khoo V, Lindeman GJ, Lubinski J, Axcrona K, Mikropoulos C, Mitra A, Moynihan C, Rennert G, Suri M, Wilson P, Dudderidge T; IMPACT Study Collaborators; Offman J, Kote-Jarai Z, Vickers A, Lilja H, Eeles RA. Interim Results from the IMPACT Study: Evidence for Prostate-specific Antigen Screening in BRCA2 Mutation Carriers. Eur Urol. 2019 Dec;76(6):831-842. doi: 10.1016/j.eururo.2019.08.019. Epub 2019 Sep 16. PMID 31537406